CLINICAL TRIAL: NCT06730958
Title: Evaluation of Serum Follistatin-Like Protein 1 Levels in Behcet's Disease and Its Association With Disease Activity
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Farrag Ahmed Mohamed, Lecturer of Rheumatology and Rehabilitation, Assiut University
Other Study IDs: SFA12024
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Behcet Syndrome
MeSH Terms: conditions — Behcet Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Behçet's disease: patients with who fulfilling the criteria for the diagnosis by International Team for the Revision of the International Criteria for Bechet's Disease
  Interventions: Diagnostic Test: serum Follistatin-like protein 1
- control group: healthy matched controls
  Interventions: Diagnostic Test: serum Follistatin-like protein 1

INTERVENTIONS:
Diagnostic Test: serum Follistatin-like protein 1 — Serum FSL1 level Test principle The kit uses a double-antibody sandwich enzyme-linked immunosorbent assay(ELISA) to assay the level ofHuman Follistatin Like Protein 1(FSTL1) in samples. Add Follistatin Like Protein 1(FSTL1)to monoclonal antibody.Enzyme well which is pre-coated with Human Follistatin Like Protein1(FSTL1)monoclonal antibody, incubation; then, add Follistatin Like Protein 1(FSTL1)antibodies labeled with biotin, and combined with Streptavidin-HRP to form immune complex; then carry out incubation and washing again to remove the uncombined enzyme. Then add Chromogen Solution A, B, the color of the liquid changes into the blue, And at the effect of acid, the color finally becomes yellow. The chroma of color and the concentration of the Human Substance Follistatin Like Protein 1(FSTL1) of sample were positively correlated.

SUMMARY:
Behçet's disease (BD) is a multi-system auto inflammatory disorder with vasculitic features.

The exact etiological of BD is still obscure, although environmental and genetics factors have been found to be involved in disease pathogenesis.FSTL-1 can act as diagnostic and prognostic biomarkers for Some inflammatory autoimmune diseases including BD.

DETAILED DESCRIPTION:
Behçet's disease (BD) is a multi-system auto inflammatory disorder with vasculitic features Clinical manifestation of BD includes recurrent oral and genital ulcerations, uveitis, skin lesions, vascular, neurological, and gastrointestinal manifestations.The exact etiological of BD is still obscure, although environmental and genetics factors have been found to be involved in disease pathogenesis.

Most of BD manifestations have features of systemic perivasculitis. Cell-mediated immunity has a significant role in BD pathogenesis . Activation of Type 1 helper T (Th1) cell will increase levels of circulating T-lymphocytes, with subsequent increase in the levels of proinflammatory cytokines accounting for most of BD symptoms. These proinflammatory cytokines may be used as an indicator of disease severity. Also Increased macrophage activation, neutrophil chemotaxis, and phagocytosis have been described in BD lesion.

Indeed, the need for studying biomarkers that may drive inflammatory pathways involved in BD pathogenesis is crucial.

Follistatin-like proteins (FLP) belong to the family of acidic cysteine-rich secreted glycoproteins (SPARC) that are highly homologous to the activin-binding protein, follistatin (FST)(7). this group of proteins include five types: FSTL1, FSTL2, FSTL3, FSTL4 and FSTL5.

Follistatin-like protein 1 (FSTL-1) is a soluble gly¬coprotein expressed by mesenchymal cells. It has been involved in various signaling pathways and biological processes. FSTL1 has dual effect in inflammatory processes and has been evaluated in some laboratory models and can serve as pro-inflammatory and anti-inflammatory markers.

During the acute inflammation FSL1 may act as an anti-inflammatory factor, while they exert a pro-inflammatory effect in chronic inflammation. This dual effect has been explained by activation of several signaling pathways.

Although, additional exogenous and endogenous factors, may be involved in such regulation. Increased serum levels FSTL1 levels were found in some of autoimmune systemic diseases including rheumatoid arthritis, Sjogren's syndrome and osteoarthritis. Moreover, the In¬creased serum levels of FSTL-1 where found to be positively correlated with disease activity in some autoim¬mune diseases, including, rheumatoid arthritis (RA), juvenile idiopathic arthritis and systemic lupus ery¬thematosus (SLE).

Based on the above mention findings, FSTL-1 can act as diagnostic and prognostic biomarkers for Some inflammatory autoimmune diseases including BD.

ELIGIBILITY:
Inclusion Criteria:

* Adult BD patients who fulfilling the criteria for the diagnosis by International Team for the Revision of the International Criteria for Bechet's Disease

Exclusion Criteria:

* Individuals with other autoimmune diseases (rheumatoid arthritis dermatomyositis, scleroderma, mixed connective tissue disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult BD patients who fulfilling the criteria for the diagnosis by International Team for the Revision of the International Criteria for Bechet's Disease
Sampling Method: Non-Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
FSL1in the serum of BD patients | 3 months
  the level of FSL1in the serum of BD patients and their relation to various disease clinical and laboratory data in addition to the correlation between FSL1 level and BD activity.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Farrag, Lecturer, Principal Investigator — Assiut University
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yazici Y, Hatemi G, Bodaghi B, Cheon JH, Suzuki N, Ambrose N, Yazici H. Behcet syndrome. Nat Rev Dis Primers. 2021 Sep 16;7(1):67. doi: 10.1038/s41572-021-00301-1. PMID 34531393
- [Result] Tortoriello DV, Sidis Y, Holtzman DA, Holmes WE, Schneyer AL. Human follistatin-related protein: a structural homologue of follistatin with nuclear localization. Endocrinology. 2001 Aug;142(8):3426-34. doi: 10.1210/endo.142.8.8319. PMID 11459787
- [Result] Kaplan H, Calis M, Yazici C, Gunturk I, Cuce I, Senel AS. Are follistatin-like protein 1 and follistatin-like protein 3 associated with inflammatory processes in patients with familial Mediterranean fever? North Clin Istanb. 2023 Jun 6;10(3):306-313. doi: 10.14744/nci.2022.54189. eCollection 2023. PMID 37435280